CLINICAL TRIAL: NCT05825768
Title: Preoperative Magnetic Resonance Imaging to Obtain Adequate Resection Margins (PRIMAR) Trial
Brief Title: Preoperative Magnetic Resonance Imaging to Obtain Adequate Resection Margins in Breast Conserving Surgery, (PRIMAR) Trial
Acronym: PRIMAR
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulties recruiting the patients at one of the sites.
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Irina Palimaru Manhoobi, Principal Investigator, Medical Doctor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NNF19OC0057928
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer
Keywords: Resection Margins; repeat surgery
MeSH Terms: conditions — Breast Neoplasms; Margins of Excision

STUDY DESIGN:
Intervention Model Description: Randomized, open-label, double-center trial including female participants with early breast cancer planned for breast conserving surgery randomised 1:1 in a Magnetic Resonance Imaging, MRI-group (preoperative MRI, ultrasound and mammography) and a control group (preoperative ultrasound and mammography).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRI-group (Active Comparator): This group of patients are allocated to a supplementary preoperative breast Magnetic Resonance Imaging (MRI) in addition to standard preoperative breast imaging (ultrasound and mammography).
  Interventions: Device: Breast MRI; Diagnostic Test: standard breast imaging
- Control group (Other): This groups of patients are allocated to receive standard preoperative breast imaging only (ultrasound and mammography).
  Interventions: Diagnostic Test: standard breast imaging

INTERVENTIONS:
Device: Breast MRI — Breast Magnetic Resonance Imaging prior to breast conserving surgery with and without intravenous contrast agent.
  Arms: MRI-group
Diagnostic Test: standard breast imaging — The control group that receives standard preoperative imaging only (breast ultrasound and mammography)

SUMMARY:
The goal of this randomised study is to investigate if a supplementary preoperative breast Magnetic Resonance Imaging (MRI) improves the assessment of breast cancer and can help surgical planning such that sufficient resection margins can be obtained during breast conserving surgery.

The main questions are:

1. Is preoperative breast MRI in addition to the currently used standard imaging methods ultrasound and mammography more accurate to detect Ductal Carcinoma in Situ and the invasive breast tumor compared to standard methods only?
2. Does preoperative breast MRI reduce the number of involved histological margins after breast conserving surgery in the MRI-group versus the control group?

DETAILED DESCRIPTION:
Magnetic Resonance Imaging (MRI) of the breast preoperatively is a well-known imaging method in primary breast cancer and is only used as a complement to the standard imaging methods in complex cases, lobular cancer, patients with large tumors that need preoperative neoadjuvant therapy or for patients with dense breast tissue where the tumor is difficult to detect with the standard imaging methods. The MRI is not used as a standard diagnostic method, because of its lower specificity that may result in a higher false-positivity rate.

The advantage of the MRI with use of intravenously contrast agent (also called dynamic enhanced MRI), is its ability to simultaneously assess the tumor morphology and semiquantitative enhancement kinetics that evaluate the newly formed vessels as a tumor-specific feature. A fast-initial enhancement and wash-out (type III) is typically seen in malignancies, due to increased vascular permeability, density, and interstitial fluid. Furthermore, the breast MRI can identify preinvasive malignant lesions such as Ductal Carcinoma in Situ (DCIS) in the breast with a much higher sensitivity than mammography and most commonly manifests as non-mass-enhanced lesion on an MRI with intravenous contrast agent. Less frequently the DCIS manifests as a mass or a focus on MRI and is usually not visible on non-contrast enhanced MRI, because it is masked by the normal breast parenchyma. Few larger randomized trials have investigated the efficacy of preoperative MRI in breast cancer and its effect on involved histological margins after breast conserving surgery that lead to repeat surgery. Controversy still exists whether preoperative MRI of the breast can reduce the number of repeat surgery in breast cancer. We aim to investigate in this randomised study if a supplementary breast MRI preoperatively with an optimised MRI scan protocol can help surgical planning to detect the DCIS and invasive cancer such that tumor free resection margins can be obtained during breast conserving surgery (BCS) and the patients can avoid repeat surgery.

Methods:

The study will be performed as a clinical, open-label, prospective and randomized study. We will include 440 breast cancer patients, randomized to either MRI of the breast prior to BCS together with the standard methods: Ultrasound and mammography (220) or to standard methods only (220) at two different breast centers, Aarhus University Hospital (AUH) and Viborg Regional Hospital (VRH).

The MRI of the breast: Will be performed with a protocol with intravenous contrast agent, Dotarem on a 3 Tesla Siemens MRI at the Department of Radiology at AUH and a 1.5 Tesla Siemens MRI System at VRH, with breast adaptive coils and diffusions sequences. The MRI of the breast will be performed soon after the patient is included in this study and will not delay surgery. The MRI protocol consists of T2- and T1-weighted spin-echo sequences in the axial plane, a T2-weighted sequence, dynamic contrast enhanced subtracted series with intravenous contrast agent Dotarem and diffusions-sequences, with breast adaptive coils at each institution. The MRI images of the breast from VRH for each patient will be sent to AUH, where the images will be interpreted by an experienced breast radiologist, using the same picture archiving and communication system from Siemens Healthcare. The tumor and DCIS will be measured, localized anatomically and presented for the breast surgeon at each institution at Multi-Disciplinary-Team conferences at each institution. The size of the invasive tumor and the DCIS in the breast will be recorded and compared to the corresponding size on the standard methods with mammography and ultrasound.

Ultrasound and mammography of the breast: Are routine methods at both institutions that are used as part of the triple diagnosis of breast cancer (palpation of the breast, ultrasound and mammography of the breast and ultrasound-guided core biopsy of the tumor). Ultrasound and mammography are performed and interpreted at both institutions by dedicated and specialized breast radiologists.

Final histopathology: The final microscopical assessment of the margins are the reference method for the final status of the margins and will be performed by experienced breast pathologists. According to the Danish Health Board´s recommendations, a final pathology report should be available after 7 workdays.

Statistical Analysis:

Power calculation: The number of repeat surgery for positive margins after BCS is in average 20%. A sample size of at least 219 patients was calculated as necessary to detect a reduction from 20% in the non-MRI group to 10% in the MRI-group with a statistical power of 80% and a 5% level of significance. We expect that few patients may drop-out for different reasons, and we estimated that a total number of 440 patients are enough to be included. Chi-square test will be used to compare outcomes with categorical variables. Regression analysis will be used for adjusted analysis. A p-value of less than 0.05 will be considered statistically significant.

Safety:

Allergic reactions to contrast intravenous contrast Dotarem with Gadolinium that we plan to use are very rare, approximately 0,1 %, where most are mild with skin rash.

Should an allergic reaction happen during contrast administration to the study patient, the radiologist will examine the patient and initiate medical treatment according to the severity of the adverse event and according to local instruction at each department. During the first consultation with the surgeon, the patient will be asked about previous allergic reactions towards contrast agents. If the patient has previously had severe allergic reaction towards the MRI contrast agent Dotarem, the patient will not be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed women with biopsy-verified invasive breast cancer
* Age > 18 year
* Eligible for Breast Conserving Surgery (BCS) based on preoperative ultrasound and mammography
* Cooperative to receive an Magnetic Resonance Imaging (MRI)-examination

Exclusion Criteria:

* Planned mastectomy
* Included patients where the planned BCS changes to mastectomy based on preoperative MRI
* Patients where a preoperative MRI is requiered (patients treated with neoadjuvant therapy and complex cases where a preoperative MRI is needed)
* Previous surgery for pre-malignant or malignant lesions in the breast
* Pregnancy and lactation
* Male breast cancer
* Contraindications for an MRI-examination (pacemaker, severe kidney insufficiency with glomerular filtration rate < 30 mL/min, and MRI incompatible implants or devices, claustrophobia, disability that prevents an MRI-examination in a prone position, allergy towards Dotarem (intravenous contrast agent for MRI)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Involved resection margins in the final histopathology | 2 weeks (Time from the day of preoperative breast Magnetic Resonance Imaging (MRI) to the final histopathology postoperatively)
  The number of involved (positive) resection margins in the final histopathology after breast conserving surgery that lead to repeat surgery.
Number of re-excisions during breast conserving surgery | 1 week
  The number of patients where additional breast tissue is removed during initial breast conserving surgery.

SECONDARY OUTCOMES:
Number of additional malignant tumors and Ductal Carcinoma in Situ (DCIS) in the breast detected | 2 weeks
  The number of additional malignant tumors and DCIS in the breast detected (MRI vs. standard methods)
Type of repeat surgery | 1
  Type of repeat surgery: Breast conserving surgery or mastectomy

CONTACTS AND LOCATIONS:
Overall Officials: Peer Christiansen, MD, DMSc, Principal Investigator — Department of Plastic- and Breast Surgery, Aarhus University Hospital
Locations (2):
- Denmark (2):
  - Department of Plastic- and Breast Surgery, Aarhus University Hospital, Aarhus
  - Department of Surgery, Viborg Regional Hospital, Viborg

IPD SHARING:
Plan to Share IPD: No
The plan is to share participant data when the inclusion ends and data analysis is final and the final manuscript is published.